CLINICAL TRIAL: NCT03365479
Title: Acute Hemodynamic Response of Iloprost Inhalation Using the Breelib Nebulizer in Pulmonary Arterial Hypertension
Brief Title: Acute Response of Iloprost Inhalation Using the Breelib Nebulizer in Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Jan Grimminger, Study Chair: Ghofrani H. Ardeschir, Prof. Dr. University of Giessen, University of Giessen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: V04_21112017
Record Dates: First submitted 2017-11-27; First posted 2017-12-07 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: pulmonary hypertension; iloprost; inhaled; breelib; nebulizer; pulmonary arterial hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Respiratory Aspiration | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study cohort (Experimental): The study comprises a 1-day Screening period, followed by a right heart catheterization with a single administration of inhaled iloprost 2.5 μg delivered via Breelib nebulizer
  Interventions: Drug: Iloprost

INTERVENTIONS:
Drug: Iloprost — Single administration of inhaled iloprost 2.5 μg delivered via Breelib nebulizer

SUMMARY:
Primary objective

• To evaluate the effect of rapid inhalation of 2.5μgiloprost using the Breelib nebulizer on pulmonary vascular resistance (PVR) in patients with pulmonary arterial hypertension

Secondary objectives

* To evaluate the effect of rapid iloprost inhalation using the Breelib nebulizer on mean pulmonary arterial pressure (mPAP), cardiac output (CO), cardiac index (CI), systemic blood pressure, arterial oxygen saturation, heart rate, and pulmonary arterial wedge pressure (PAWP).
* To evaluate the safety and tolerability of the rapid iloprost inhalation using the Breelib nebulizer.

DETAILED DESCRIPTION:
This study aims to investigate the acute hemodynamic and pharmacological effects of a single inhalation of Iloprost (2.5μg) during right heart catheterization (RHC) using the Breelib nebulizer. Patients with confirmed diagnosis of pulmonary arterial hypertension (PAH = WHO group 1), NYHA functional class III and with stable background pulmonary vasoactive treatment or treatment naïve PAH patients will be challenged with the iloprost inhalation dosage during RHC. As a proof-of concept design, the study will include consecutive PAH patients only challenged with a single administration of inhaled iloprost 2.5 μg delivered via Breelib nebulizer during right heart catheterization (day 2).

The acute hemodynamic response will be followed over 30 minutes. Change of pulmonary hemodynamics, systemic blood pressure, right ventricular echocardiographic parameters and adverse events will be assessed at baseline and 5, 10, 15, 30 minutes after the end of inhalation.

Recently, the Breelib nebulizer has been evaluated within a multicenter, randomized, unblinded, study. This safety and feasibility study compared inhalation time, pharmacokinetics, and acute tolerability of inhaled iloprost delivered via Breelib versus the standard I-Neb nebulizer. The primary safety endpoints (AEs) were reported with a low frequency and were consistent with the known safety profile of iloprost. Median inhalation times were considerably shorter while maximum iloprost plasma concentration and systemic exposure were significantly higher, with Breelib versus I-Neb. Previously, it was shown that the acute hemodynamic response of iloprost inhalation via the previous used I-Neb nebulizer resulted in a relevant and significant reduction of PVR and increase in CI. Moreover, previous generation of nebulizers also resulted in a significant reduction of PVR and increase in CI 5-15min after iloprost inhalation.

Therefore, the aim of the current study is to determine the acute hemodynamic effects on the pulmonary and the systemic circulation as well as on the gas exchange of 2.5 μg iloprost delivered via the Breelib device. The investigators aim to characterize the hemodynamic profile of the inhalation with Breelib as the investigators speculate that the shortened inhalation time will result in an enhanced hemodynamic response with substantial reduction of pulmonary vascular resistance (PVR). Moreover, as a secondary outcome measurement the investigators aim to assess the response of mean pulmonary arterial pressure, cardiac index/cardiac output, systemic blood pressure, right ventricular echocardiographic parameters and oxygen saturation after inhalation of 2.5μg iloprost and analyze adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pulmonary arterial hypertension, WHO group 1 diagnosed according to current guidelines
* New York Heart Association functional class III
* mPAP ≥ 25 mmHg, PAWP ≤ 15 mmHg
* Age ≥ 18 years; ≤ 85 years
* planned right heart catheterization based on clinical grounds
* Stable specific PAH medications other than prostanoids
* Signed informed consent

Exclusion Criteria:

* other etiologic groups of pulmonary hypertension (WHO group 2, 3, 4, 5)
* Unstable or severe coronary artery disease (history of cardiac surgery, history of coronary intervention 2 years prior to inclusion), uncontrolled arterial hypertension, severe left ventricular hypertrophy, severe congenital or acquired valvular or myocardial disease, systolic blood pressure < 90 mmHg, heart rate of <55 or >105 beats·min-1 before inhalation
* Progressive left heart failure History of severe ventricular arrhythmias
* Pulmonary veno-occlusive disease
* Transitory ischemic attack (TIA) or stroke ≤ 3months
* Severe hepatic impairment (> CHILD B)
* Severe, terminal renal impairment
* Use of intravenous, subcutaneous or oral prostacyclin/IP receptor agonists
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Change of PVR (∆PVR) | 5, 10, 15, 30 minutes after the end of inhalation

SECONDARY OUTCOMES:
Change of mPAP | at baseline and 5, 10, 15, 30 minutes after the end of inhalation
Change of PAWP | at baseline and 5, 10, 15, 30 minutes after the end of inhalation
Change of CI | at baseline and 5, 10, 15, 30 minutes after the end of inhalation
Change of systemic blood pressure | 5, 10, 15, 30 minutes after the end of inhalation
Change of oxygen saturation | 5, 10, 15, 30 minutes after the end of inhalation
Change of right heart echocardiography | 5, 10, 15, 30 minutes after the end of inhalation
Adverse events (AEs) | 5, 10, 15, 30 minutes after the end of inhalation

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Clinic Giessen and Marburg, Giessen, Hesse
  - Kerckhoff-Klinik, Bad Nauheim

IPD SHARING:
Plan to Share IPD: No